CLINICAL TRIAL: NCT03720119
Title: Multicentre Observational Study on the Wound Pain Relief Properties of ORTODERMINA®
Status: Completed | Type: Observational
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: SINALGO
Record Dates: First submitted 2018-10-15; First posted 2018-10-25 (Actual); Results first posted 2019-11-07 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2019-10

CONDITIONS: Wound Healing Disorder
Keywords: wound healing; pain; lidocaine
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — As per clinical practice, a local treatment with ORTODERMINA® over a 14-day period (once a day) was prescribed. ORTODERMINA® contains 5% of lidocaine hydrochloride.
  Other Names: ORTODERMINA®

SUMMARY:
Acute pain may occur due to trauma, surgery, infection, disruption of blood circulation or when there is tissue injury. It can be managed using analgesics and conduction anaesthesia, which may be preferable because of superior pain control and fewer side effects. Lidocaine hydrochloride is used topically to relieve itching, burning and pain from skin inflammation. This multicentric observational study is aimed to evaluate the relief gained with lidocaine hydrochloride (ORTODERMINA®) on wound pain in patients with painful wounds and to collect safety information on this treatment.

DETAILED DESCRIPTION:
Acute pain can be managed using analgesics and conduction anaesthesia which may be preferable because of superior pain control and fewer side effects. In this contest, lidocaine hydrochloride (ORTODERMINA®) plays an important role in pain management during wound healing. The properties of ORTODERMINA® and its ability to maintain an adequate level of active drug over the lesion allow a persistent anaesthetic effect. ORTODERMINA® is a drug for topical application in the form of cream, with a high safety profile. However, although the incidence of adverse effects with Lidocaine Ointment 5% is quite low, caution should be exercised, particularly when employing large amounts, since the incidence of adverse effects is directly proportional to the total dose of local anaesthetic agent administered.

This multicentric observational study is aimed to evaluate the relief gained with ORTODERMINA® on wound pain in patients with painful wounds and to collect safety information on this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients with painful exuding wounds >1 cm2 that includes painful exuding ulcers and pressure ulcers grade II [according to National Pressure Ulcer Advisory Panel (NPUAP) classification]
* Patients available and able to return to the study site for the scheduled visits
* Patients who gave written informed consent to take part into the study

Exclusion Criteria:

* Patients with ulcer infected, discoloured, odorous, pressure ulcer grade I, III, or IV (according to NPUAP classification)
* Diabetic foot ulcer
* Patients with contraindication or known allergy to drug's components
* Patients with known severe allergies manifested by a history of anaphylaxis, or history or presence of severe multiple allergies
* Patients who are pregnant or lactating.
* Patients with vascular disorders (mainly arteriopathies)
* Patients known as alcohol or drug abusers.
* Patients currently participating in a clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample size of 70 evaluable patients is needed to test the hypothesis of an improvement in wound pain relief and a reduction in pain intensity, assuming a standardized effect size equal to 0.35, for a one-tailed test with a 5% significance level and a 90% power. A 10% of attrition rate is expected; therefore, a total number of patients to be enrolled is 78.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Romanelli, MD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana; Elia Ricci, MD, Study Chair — Clinica San Luca, Torino
Locations (2):
- Italy (2):
  - Azienda Ospedaliero Pisana, Pisa
  - Ospedali Riuniti Trieste, Trieste

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips TJ. Chronic cutaneous ulcers: etiology and epidemiology. J Invest Dermatol. 1994 Jun;102(6):38S-41S. doi: 10.1111/1523-1747.ep12388556. PMID 8006433
- [Background] Dallam L, Smyth C, Jackson BS, Krinsky R, O'Dell C, Rooney J, Badillo C, Amella E, Ferrara L, Freeman K. Pressure ulcer pain: assessment and quantification. J Wound Ostomy Continence Nurs. 1995 Sep;22(5):211-5; discussion 217-8. doi: 10.1097/00152192-199509000-00007. PMID 7550776
- [Background] Vandenkerkhof EG, Hopman WM, Carley ME, Kuhnke JL, Harrison MB. Leg ulcer nursing care in the community: a prospective cohort study of the symptom of pain. BMC Nurs. 2013 Feb 6;12:3. doi: 10.1186/1472-6955-12-3. PMID 23388350
- [Background] Chase SK, Melloni M, Savage A. A forever healing: the lived experience of venous ulcer disease. J Vasc Nurs. 1997 Jun;15(2):73-8. doi: 10.1016/s1062-0303(97)90004-2. PMID 9238945
- [Background] Briggs M, Closs SJ. Patients' perceptions of the impact of treatments and products on their experience of leg ulcer pain. J Wound Care. 2006 Sep;15(8):333-7. doi: 10.12968/jowc.2006.15.8.26941. PMID 17001939
- [Background] Khaliq W, Alam S, Puri N. Topical lidocaine for the treatment of postherpetic neuralgia. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004846. doi: 10.1002/14651858.CD004846.pub2. PMID 17443559
- [Background] Santiago S, Ferrer T, Espinosa ML. Neurophysiological studies of thin myelinated (A delta) and unmyelinated (C) fibers: application to peripheral neuropathies. Neurophysiol Clin. 2000 Feb;30(1):27-42. doi: 10.1016/S0987-7053(00)88865-6. PMID 10740794
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Pocock SJ. Clinical trials with multiple outcomes: a statistical perspective on their design, analysis, and interpretation. Control Clin Trials. 1997 Dec;18(6):530-45; discussion 546-9. doi: 10.1016/s0197-2456(97)00008-1. PMID 9408716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from January 27, 2015 to March 05, 2018 in three Italian hospitals in Pisa and Trieste
Groups:
- Single Cohort: A single cohort of 78 patients with painful wounds >1 cm2 -painful ulcers and pressure ulcers grade II, per NPUAP classification-, both sexes, aged ≥18 years. Patients were treated with Ortodermina, as per clinical practice. Three investigational sites have been involved.
Period: Overall Study
Arm/Group | Single Cohort
Started | 78
Completed | 69
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Single Cohort
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (21.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 78
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Type of wounds [Count of Participants; unit: Participants]
  Traumatic | 39
  Pathological | 31
  Surgical | 7
  Geriatric | 1
Size of wounds [Mean (Standard Deviation); unit: cm]
  Width | 5.99 (5.13)
  Length | 4.76 (3.35)
  Depth | 0.29 (0.29)
Presence of exudate [Count of Participants; unit: Participants]
  Present | 53
  Not present | 23
  Not defined | 2
Odour of wounds [Count of Participants; unit: Participants]
  Absent | 78
  Present | 0
Edges of wounds [Count of Participants; unit: Participants]
  Regular | 40
  Irregular | 18
  Reactive | 11
  Herythematous | 6
  Not defined | 3
Colour of wounds [Count of Participants; unit: Participants]
  Pink/red/yellow | 68
  Not defined | 10
Wounds classification [Count of Participants; unit: Participants] — Definition of NPUAP Stage 2 Pressure Injury: Partial-thickness skin loss with exposed dermis
  Participants
    NPUAP Grade II | 60
    Not available | 18
Concomitant Therapies [Count of Participants; unit: Participants]
  1 therapy | 19
  2-4 therapies | 25
  >4 therapies | 6
  No therapy | 28

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain Relief From Baseline to the End of Treatment Using the 5-point Visual Rating Scale (VRS)
Description: The evaluation of wound pain relief was based on a 5-point Visual Rating Scale (0 = none improvement; 4 = total relief).
  Patients recorded the VRS score every day of treatment in their diary. The improvement in the pain relief was defined as a VRS scores at end of treatment significantly greater than 0.
Time Frame: Every day for 15 days
Population: There are missing data in some time-points
Measure: Count of Participants; unit: Participants
Arm/Group | Single Cohort
Number analyzed (Participants) | 78
Participants
  Day 2: number analyzed (Participants) | 77
  Day 2: None relief | 3
  Day 2: Mild | 23
  Day 2: Moderate | 28
  Day 2: A lot | 20
  Day 2: Complete relief | 3
  Day 3: number analyzed (Participants) | 76
  Day 3: None relief | 2
  Day 3: Mild | 24
  Day 3: Moderate | 30
  Day 3: A lot | 18
  Day 3: Complete relief | 2
  Day 4: number analyzed (Participants) | 77
  Day 4: None relief | 3
  Day 4: Mild | 24
  Day 4: Moderate | 31
  Day 4: A lot | 15
  Day 4: Complete relief | 4
  Day 5: number analyzed (Participants) | 76
  Day 5: None relief | 5
  Day 5: Mild | 17
  Day 5: Moderate | 39
  Day 5: A lot | 11
  Day 5: Complete relief | 4
  Day 6: number analyzed (Participants) | 73
  Day 6: None relief | 6
  Day 6: Mild | 21
  Day 6: Moderate | 33
  Day 6: A lot | 9
  Day 6: Complete relief | 4
  Day 7: number analyzed (Participants) | 70
  Day 7: None relief | 5
  Day 7: Mild | 16
  Day 7: Moderate | 35
  Day 7: A lot | 9
  Day 7: Complete relief | 5
  Day 8: number analyzed (Participants) | 70
  Day 8: None relief | 7
  Day 8: Mild | 18
  Day 8: Moderate | 25
  Day 8: A lot | 15
  Day 8: Complete relief | 5
  Day 9: number analyzed (Participants) | 66
  Day 9: None relief | 5
  Day 9: Mild | 22
  Day 9: Moderate | 22
  Day 9: A lot | 14
  Day 9: Complete relief | 3
  Day 10: number analyzed (Participants) | 67
  Day 10: None relief | 10
  Day 10: Mild | 16
  Day 10: Moderate | 22
  Day 10: A lot | 16
  Day 10: Complete relief | 3
  Day 11: number analyzed (Participants) | 64
  Day 11: None relief | 10
  Day 11: Mild | 16
  Day 11: Moderate | 20
  Day 11: A lot | 14
  Day 11: Complete relief | 4
  Day 12: number analyzed (Participants) | 65
  Day 12: None relief | 12
  Day 12: Mild | 14
  Day 12: Moderate | 20
  Day 12: A lot | 14
  Day 12: Complete relief | 5
  Day 13: number analyzed (Participants) | 64
  Day 13: None relief | 16
  Day 13: Mild | 10
  Day 13: Moderate | 20
  Day 13: A lot | 14
  Day 13: Complete relief | 4
  Day 14: number analyzed (Participants) | 60
  Day 14: None relief | 14
  Day 14: Mild | 11
  Day 14: Moderate | 20
  Day 14: A lot | 12
  Day 14: Complete relief | 3
  Day 15: number analyzed (Participants) | 58
  Day 15: None relief | 13
  Day 15: Mild | 13
  Day 15: Moderate | 15
  Day 15: A lot | 13
  Day 15: Complete relief | 4

2. Primary Outcome: Change of Pain Intensity From Baseline to the End of Treatment Using the 11-point Numerical Pain Rating Scale (NPRS)
Description: The evaluation of the pain intensity was based on a 11-point Numerical Pain Rating Scale (NPRS score from 0= no pain to 10= the most intense pain imaginable). Patients recorded the NPRS score every day of treatment in their diary.
  The improvement in the pain intensity is defined as a decrease in NPRS scores from baseline to the end of treatment.
Time Frame: Every day for 15 days
Population: The degree of pain intensity was recorded by patients on daily diary and revised by Investigators at final visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Single Cohort
Number analyzed (Participants) | 78
Score on a scale
  NPRS score of Day 1 | 6.7 (1.90)
  NPRS score of Day 2 | 5.4 (1.91)
  NPRS score of Day 3: number analyzed (Participants) | 77
  NPRS score of Day 3 | 5.0 (2.09)
  NPRS score of Day 4: number analyzed (Participants) | 77
  NPRS score of Day 4 | 4.7 (2.17)
  NPRS score of Day 5: number analyzed (Participants) | 76
  NPRS score of Day 5 | 4.1 (2.16)
  NPRS score of Day 6: number analyzed (Participants) | 73
  NPRS score of Day 6 | 3.9 (2.2)
  NPRS score of Day 7: number analyzed (Participants) | 70
  NPRS score of Day 7 | 3.6 (2.05)
  NPRS score of Day 8: number analyzed (Participants) | 70
  NPRS score of Day 8 | 3.6 (2.22)
  NPRS score of Day 9: number analyzed (Participants) | 66
  NPRS score of Day 9 | 3.6 (2.22)
  NPRS score of Day 10: number analyzed (Participants) | 67
  NPRS score of Day 10 | 3.4 (2.28)
  NPRS score of Day 11: number analyzed (Participants) | 63
  NPRS score of Day 11 | 3.2 (2.40)
  NPRS score of Day 12: number analyzed (Participants) | 65
  NPRS score of Day 12 | 3.2 (2.40)
  NPRS score of Day 13: number analyzed (Participants) | 64
  NPRS score of Day 13 | 3.3 (2.48)
  NPRS score of Day 14: number analyzed (Participants) | 59
  NPRS score of Day 14 | 3.0 (2.27)
  NPRS score of Day 15: number analyzed (Participants) | 58
  NPRS score of Day 15 | 2.8 (2.23)
Statistical Analysis 1: Comparison: Single Cohort; Test type: Other — Analysis of Variance for repeated measurements; p = 0.0001, Dunnett's post-hoc test — The calculated P-Value represents the repeated measurement/Day (all times versus Day 1); day effect F = 27.83

3. Secondary Outcome: Incidence and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Evaluation of incidence and severity of AEs and SAEs in all patients entered in the study
Time Frame: 15 days, starting from informed consent signature up to the end of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Single Cohort
Number analyzed (Participants) | 78
Participants
  0 adverse event | 65
  1 adverse event | 8
  2 adverse events | 1
  3 adverse events | 2
  4 adverse events | 1
  5 adverse events | 1

ADVERSE EVENTS:
Time Frame: 15 days, from informed consent signature to the end of the study
Arm/Group | Single Cohort
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 13/78
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Cohort (N=78)
Pain (Musculoskeletal and connective tissue disorders) | 3 (6) — Pain Lower part of the Leg
Infection (Infections and infestations) | 3 (4)
BURNING SENSATION (Injury, poisoning and procedural complications) | 1 (4)
Stomach Ache (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 3 (3)
PYODERMA GANGRENOSUM (Infections and infestations) | 1 (1)
COUGH (Infections and infestations) | 1 (2)
ACCIDENTAL FALL WITH FACIAL TRAUMA (Injury, poisoning and procedural complications) | 1 (1)
FEVER (General disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Wound Pain (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
There are not limitations or caveats to be reported for this clinical investigation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT03720119/Prot_SAP_000.pdf